CLINICAL TRIAL: NCT02196883
Title: A Prospective, Randomized, Single Blind Study Comparing Transforaminal Epidural Steroid Injections at the Level of MRI Pathology vs Clinical Symptoms
Brief Title: Steroid Injections Given at the "Level of MRI Pathology" Versus at the "Level of Clinical Symptoms" to See if One is More Effective Than the Other.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI no longer part of practice
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 593154-1
Record Dates: First submitted 2014-07-18; First posted 2014-07-22 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2014-07

CONDITIONS: Radiculopathy; Spinal Stenosis; Intervertebral Disc Displacement
MeSH Terms: conditions — Radiculopathy; Spinal Stenosis; Intervertebral Disc Displacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MRI Pathology (Active Comparator)
  Interventions: Procedure: Transforaminal Epidural Steroid Injection
- Physical Exam Pathology (Active Comparator)
  Interventions: Procedure: Transforaminal Epidural Steroid Injection

INTERVENTIONS:
Procedure: Transforaminal Epidural Steroid Injection

SUMMARY:
Patients are being asked to participate in a research study because the patients are being treated for low back pain and the patients have decided to have an epidural steroid injection.

Low back pain has a tremendous impact on the individual and society. It not only affects the individuals quality of life, it also contributes to lost productivity and increased health care costs.

Epidural steroid injections (ESIs) are a common treatment option for many forms of low back pain. They have been used for low back problems since 1952 and are still being used as a non-surgical form of treatment for low back pain. The goal of the injections is reduction of pain, increased quality of life and improved function.

This study is being conducted to determine the outcomes of injections given at the "level of MRI Pathology" versus at the "level of clinical symptoms" to see if one is more effective than the other and to learn more about the characteristics of the two different injections.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Single level spinal stenosis.
* Single level radiculopathy with MRI findings at a different level than clinical pattern.
* Chronic low back pain with radicular symptoms of > 4 weeks, but < 6 months.
* Failure of conservative therapy to include physical and pharmacotherapy.
* Patient is at least 21 years of age.
* Patient is willing to be blinded to treatment until after the 3-month follow up visit.
* Patient is willing and able to review and sign the study's informed consent form.

Exclusion Criteria:

* Patient has a mental or physical condition that would invalidate evaluation results.
* Patient has had prior lumbar surgery at any level.
* Patient is pregnant.
* Patient has systemic infection or infection at the proposed injection site.

Min Age: 21 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-05; Primary Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | 2 weeks to 6months

SECONDARY OUTCOMES:
Short Form 36 Health Survey | 2 weeks to 6months
Oswestry Disability Index | 2 weeks to 6months

CONTACTS AND LOCATIONS:
Locations (1):
- SUNY Upstate Medical Center, Syracuse, New York, United States